CLINICAL TRIAL: NCT02773108
Title: Somatic Comorbidities in Psychiatric Patients
Acronym: SCPP
Status: Completed | Type: Observational
Sponsor: Sveti Ivan Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Ena Ivezic, MA, Sveti Ivan Psychiatric Hospital
Other Study IDs: komorbiditeti
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia; Major Depression Disorder; Bipolar Affective Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hospitalized: Hospitalized psychiatric patients
- Daily hospital
- Outpatients

SUMMARY:
Prevalence of somatic comorbidities in psychiatric patients hospitalized in Psychiatric hospital or treated ambulatory or in daily hospital. Comparison of prevalence of somatic comorbidities in psychiatric patients population and the general Croatian population.

ELIGIBILITY:
Inclusion Criteria:

* treatment in psychiatric hospital

Exclusion Criteria:

* acute suicidality
* dementia
* mental retardation
* acute psychosis
* intoxication
* inability to answer the questionnaire by themselves

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients
Sampling Method: Non-Probability Sample
Enrollment: 1061 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of somatic comorbidities | 12 months

SECONDARY OUTCOMES:
Clinical Global Impression- Improvement scale (CGI-I), Change from diagnosis | from baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- PB Sveti Ivan, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jelec V, Bajic Z, Simunovic Filipcic I, Portolan Pajic I, Sentija Knezevic M, Miloloza I, Radic-Kristo D, Benjak T, Jaksic N, Sagud M, Wang W, Filipcic I. Utilization of somatic healthcare in Croatian patients with schizophrenia spectrum disorder, major depression, PTSD and the general population. BMC Psychiatry. 2019 Jun 28;19(1):203. doi: 10.1186/s12888-019-2190-8. PMID 31253196